CLINICAL TRIAL: NCT04930627
Title: Evaluation of Efficacy and Safety of Empagliflozin in Treatment of Neutropenia in Patients With Glycogenosis Ib
Brief Title: Safety and Efficacy of Empagliflozin in GSD1b Patients With Neutropenia
Acronym: EMPAtia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Department of Internal Medicine, Hypertension and Vascular Diseases, The Medical University of Warsaw (Unknown)
Responsible Party: Principal Investigator, Dariusz Rokicki, Pricipal Investigator, Children's Memorial Health Institute, Poland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMPAtia; 2021-000580-78 (EudraCT Number)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Glucose 6 Phosphatase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type I | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- oral administration of Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — dosis depending on body weight: <20 kg 5 mg 1x/day; 20-40 kg 2 x 5 mg; >40 kg 2 x 10 mg
  Other Names: Jardiance

SUMMARY:
Treatment of neutropenia of Glycogenosis type 1b patients with empagliflozin

DETAILED DESCRIPTION:
Symptoms of glycogen storage disease type Ib (GSD Ib) include - among others - hypoglycemia, hepatomegaly and neutropenia with concomitant neutrophil dysfunction, which results in recurrent bacterial and fungal infections, and inflammatory bowel disease.

At present filgrastim is the only available drug to treat neutropenia in GSD Ib patients; it stimulates neutrophil production, but doesn't restore their function. Part of GSD Ib patients doesn't respond to filgrastim treatment. The latest research results showed, that neutropenia and neutrophil dysfunction in GSD Ib patients are results of extensive accumulation of 1,5-anhydroglucitol-phosphate. Empagliflozin, a SGLT2 inhibitor, inhibits renal glucose and 1,5-anhydroglucitol reabsorption and is an effective and safe method of treatment of neutropenia in this group of patients. Empagliflozin (Jardiance®) is a drug, which is registered in Poland to treat type II diabetes in adults. The aim of our study is to evaluate the efficacy and safety of neutropenia in patients with GSD Ib with empagliflozin (Jardiance®).

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 4 weeks old female Or Male
* GSD1b confirmed by genetic analysis with neutropenia and/or reduced respiratory burst
* Informed consent signed by the parents/assigns, and the recipient (>13 years old)

Exclusion Criteria:

* Risk of non-compliance
* Chronic renal diseases (eGFR < 60 ml/min/1,73 m2)
* Active urinary tract infection (temporal criterion, up to recovery)
* Participation in another clinical trial (minimum 6 months from the end of participation until the date of signing the Informed Consent Form)
* Participation in therapeutic experiment, in addition to the experimental treatment with empagliflozin (minimum 12 months from the end of participation until the date of signing the Informed Consent Form)
* Pregnancy, breastfeeding
* Allergy to Empagliflozin
* Lack of informed consent

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Empaglifozin safety and tolerability measured by occurrence of adverse reactions | 2 years
  Empaglifozin saftey and tolerability measured by occurrence of adverse reactions

SECONDARY OUTCOMES:
Efficacy of neutropenia treatment measured as percentage of the patients | 2 years
  who achieved >500 neutrophils/ml for at least 6 months with normalization of oxidative burst with decrease of bacterial and fungal infections compared to the period before study with decrease of hospitalization number with decrease of the number of defecation, gingival sores, and calprotectin average concentration in stool
Dosis change/withdrawal of filgrastrim | 2 years
  Dosis change/withdrawal of filgrastrim
Degree of metabolic compensation | 2 years
  measured as change of triglycerides (mg/dL), lactate (mg/dL), and uric acid (mg/dL) compared to the period before study

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Memorial Health Institute, Warsaw, Poland